CLINICAL TRIAL: NCT02587975
Title: Pharmacodynamics Study to Investigate the Effect of Evogliptin on Bone Metabolism in Healthy Volunteers
Brief Title: Effect of Evogliptin on Bone Metabolism in Human
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Namyi Gu, Assistant professor, DongGuk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DUMC-EVOG-BONE
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus, Type 2; Osteoporosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Osteoporosis | interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evogliptin 10 mg (Experimental): Single oral administration of 2 tablets of evogliptin 5 mg with water 250 mL
  Interventions: Drug: Evogliptin

INTERVENTIONS:
Drug: Evogliptin — 10 mg
  Other Names: DA-1229; Suganon

SUMMARY:
This study is designed to measure the effect of evogliptin on bone metabolism in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal healthy women (at least 5 years)
* BMI 18~30 kg/m2

Exclusion Criteria:

* Presence or history of hypersensitivity or allergic reactions to any drug
* Clinically relevant abnormal medical history or present disease
* Presence or history of drug abuse
* Participation in other clinical trial within 2 months before dose.
* Bood donation during 2 months or apheresis during 1 month before the study.
* Use of a prescription medicine, herbal medicine within 2 weeks or over-the-counter medication or vitamin substances within 1 week before dose.
* Use of any drug which can affect bone metabolism such as sex hormones or their receptor related medicine, calcitonin or parathyroid hormone related medicine, systemic corticosteroid, bisphosphate, or etc.
* Smoking of more than 10 cigarettes/days within 3 months before first dose.
* Use of alcohol over 21 units/weeks
* Subject judged not eligible for study participation by investigator.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-11 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Serum concentration of C-terminal telopeptide after treatment in comparison with the baseline | Predose and 1, 2, 3, 4, 6, 14, 20, 24 h postdose on Day 1 and Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Namyi Gu, MD, PhD, Principal Investigator — Dongguk University College of Medicine and Ilsan Hospital
Locations (1):
- Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea